CLINICAL TRIAL: NCT00002949
Title: Phase I Study of Concomitant Chemoradiotherapy With Vinorelbine and Paclitaxel in Patients With Advanced Pelvic Malignancies
Brief Title: Vinorelbine and Paclitaxel Plus Radiation Therapy in Treating Patients With Advanced Cancer Arising in the Pelvis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8270; UCCRC-8270; NCI-G97-1156
Record Dates: First submitted 1999-11-01; First posted 2004-06-16 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Bladder Cancer; Cervical Cancer; Endometrial Cancer; Vaginal Cancer
Keywords: stage II cervical cancer; stage III cervical cancer; stage IV cervical cancer; stage II vaginal cancer; stage III vaginal cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; stage II endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Vaginal Neoplasms | interventions — Paclitaxel; Vinorelbine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Vinorelbine (qwk, 10, 15, 20 or 25 mg/m2), Radiation therapy (Total pelvic RT of 45 Gy in 1.8-Gy daily fractions, 85 Gy in cervical cancer patients using intracavitary brachytherapy, 70 Gy in patients treated with interstitial brachytherapy) Paclitaxel (qwk, starting dose of 20mg/m2 with planned dose escalation increments of 5mg/m2)
  Interventions: Drug: paclitaxel; Drug: vinorelbine tartrate; Radiation: radiation therapy

INTERVENTIONS:
Drug: paclitaxel — Paclitaxel (qwk, starting dose of 20mg/m2 with planned dose escalation increments of 5mg/m2)
Drug: vinorelbine tartrate — Vinorelbine (qwk, 10, 15, 20 or 25 mg/m2),
Radiation: radiation therapy — Radiation therapy (Total pelvic RT of 45 Gy in 1.8-Gy daily fractions, 85 Gy in cervical cancer patients using intracavitary brachytherapy, 70 Gy in patients treated with interstitial brachytherapy)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy with may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of chemotherapy with vinorelbine and paclitaxel plus radiation therapy in treating patients with advanced cancer arising in the pelvis.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxic effects of vinorelbine given on a weekly schedule combined with standard whole pelvic radiation therapy. II. Determine the Maximum Tolerated Dose (MTD) of vinorelbine given on a weekly schedule combined with standard whole pelvic radiation therapy. III. Access the toxic effects of paclitaxel given weekly in combination with the regimen determined to be the MTD of vinorelbine. IV. Determine the MTD of paclitaxel given weekly in combination with the regimen determined to be the MTD of vinorelbine.

OUTLINE: Part I: Vinorelbine IV bolus is administered over 8-10 minutes on day 1 prior to radiation therapy. Whole pelvic radiation treatment is given on days 1-5 followed by 2 days of rest. The treatment volume encompasses all suspected pelvic disease with a minimum of 1 cm margin. Cycles repeat weekly. Dose of vinorelbine is escalated in cohorts of at least 3 patients until maximum tolerated dose (MTD) is determined. Part II: Paclitaxel is infused over 1 hour immediately following vinorelbine at the MTD, as determined in part I. Dose of paclitaxel is escalated in cohorts of at least 3 patients until the MTD is determined. At least 6 patients are treated at the MTD for both parts I and II of the study. Patients are followed for late and chronic toxicities.

PROJECTED ACCRUAL: Projected accrual is 12 patients per year for approximately 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed locally advanced carcinoma of the uterine cervix, vagina, or bladder or other pelvic malignancy for which whole pelvic radiation therapy is planned Metastatic disease is permitted

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: CALGB 0-2 Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin within normal limits Renal: Creatinine no greater than 2.5 mg/dL Cardiovascular: No unstable angina or myocardial infarction in previous 6 months Other: Not pregnant No significant concomitant illness, uncontrolled infection, or cirrhosis

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior whole pelvic radiation therapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 1996-07; Primary Completion 2000-11 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Gini F. Fleming, MD, Study Chair — University of Chicago
Locations (1):
- University of Chicago Cancer Research Center, Chicago, Illinois, United States